CLINICAL TRIAL: NCT00096200
Title: A Phase II Trial Of BAY 43-9006, A Novel Raf Kinase Inhibitor Plus Paclitaxel/Carboplatin In Women With Recurrent Platinum Sensitive Epithelial Ovarian, Peritoneal Or Fallopian Tube Cancer
Brief Title: Sorafenib With or Without Paclitaxel and Carboplatin in Treating Patients With Recurrent Ovarian Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00067; NCI-2009-00067 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 2804; CDR0000390331; CASE 2804 (Other: Case Comprehensive Cancer Center); 6557 (Other: CTEP); N01CM62208 (NIH); P30CA043703 (NIH); U01CA062502 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; Sorafenib

ARMS (2):
- Arm I (closed to accrual 10/10/2008) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression crossover to arm II
  Interventions: Drug: Sorafenib Tosylate
- Arm II (Experimental): Patients receive oral sorafenib twice daily on days 2-19. Patients also receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Sorafenib Tosylate

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II
Drug: Sorafenib Tosylate — Given orally
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
Sorafenib may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving sorafenib together with chemotherapy may kill more tumor cells. This randomized phase II trial is studying how well giving sorafenib together with paclitaxel and carboplatin works in treating patients with recurrent ovarian cancer, primary peritoneal cancer, or fallopian tube cancer. (Sorafenib only group closed as of 10/10/2008).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES :

I. Compare the progression-free and overall survival rate of patients with recurrent platinum-sensitive ovarian epithelial, primary peritoneal, or fallopian tube cancer treated with sorafenib with or without carboplatin and paclitaxel. (Arm I [sorafenib only] closed to accrual 10/01/2008) II. Evaluate the response rate and time to disease progression in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to performance status and participating center.

ARM I (closed to accrual 10/01/2008): Patients receive oral sorafenib twice daily on days 1-28.Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression crossover to arm II.

ARM II: Patients receive oral sorafenib twice daily on days 2-19. Patients also receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian epithelial, primary peritoneal, or fallopian tube cancer
* Recurrent disease
* Must have received a prior platinum-based regimen
* Platinum-sensitive (treatment-free interval > 6 months)
* No more than 2 prior chemotherapy regimens
* Measurable disease
* At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Not in a prior irradiation field
* No known brain metastases
* Performance status:

  * ECOG 0-2 OR
  * Karnofsky 80-100%
* Life expectancy:

  * More than 12 weeks
* Hematopoietic:

  * Absolute neutrophil count >= 1,500/mm3
  * Platelet count >= 100,000/mm3
  * Hemoglobin >= 9 g/dL
  * No bleeding diathesis
* Hepatic:

  * Bilirubin < 1.5 times upper limit of normal (ULN)
  * AST or ALT =< 2 times ULN
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to sorafenib or other agents used in the study
* Patients who have had a reaction to a taxane or a platinum and have not yet been rechallenged may undergo a desensitization regimen on study
* No hypersensitivity to paclitaxel or drugs using the vehicle Cremophor El:
* Prior hypersensitivity reaction to paclitaxel allowed provided rechallenged successfully
* Renal:

  * Creatinine < 2 mg/dL
* Cardiovascular:

  * Abnormal cardiac conduction (e.g., bundle branch block or heart block) allowed if stable for the past 6 months
  * No symptomatic congestive heart failure
  * No uncontrolled hypertension
  * No cardiac arrhythmia
  * No unstable angina pectoris;
  * No myocardial infarction within the past 6 months
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate intestinal function
* No concurrent requirements for IV hydration or nutritional support
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* No other invasive malignancy with the past 5 years except nonmelanoma skin cancer
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* More than 3 weeks since prior hormonal therapy
* More than 4 weeks since prior radiotherapy and recovered
* No prior sorafenib
* No prior anticancer therapy that contraindicates study therapy
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, or phenobarbital), rifampin, or Hypericum perforatum (St. John's wort)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic anticoagulation therapy
* Concurrent prophylactic low-dose warfarin allowed for maintenance of venous or arterial access devices
* No other concurrent anticancer therapies
* No other concurrent investigational agents
* Not pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-08; Primary Completion 2011-04-21 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Waggoner, Principal Investigator — Case Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Moffitt Cancer Center at Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Case Western Reserve University, Cleveland, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients accrued from medical clinic from August 2004 through June 2011
Groups:
- Arm A: Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression crossover to arm II
- Arm B: Patients receive oral sorafenib twice daily on days 2-19. Patients also receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm C: Patients from Arm A that had progressive disease were eligible to crossover to Arm B
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 9 | 30 | 5
Completed | 8 | 23 | 5
Not Completed | 1 | 7 | 0
Not completed — Adverse Event | 0 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Ineligible pathology | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 9 | 30 | 5 | 44
Age, Customized [Number; unit: participants] — Age in years
  participants
    Age 40-49 | 0 | 2 | 0 | 2
    Age 50-59 | 4 | 15 | 0 | 19
    Age 60-69 | 4 | 8 | 5 | 17
    Age 70-79 | 1 | 5 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 30 | 5 | 44
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 22 | 5 | 35
  Unknown or Not Reported | 1 | 8 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 24 | 5 | 38
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 9 | 30 | 5 | 44

OUTCOME MEASURES:

1. Primary Outcome: Complete and Partial Response Rate Using the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Patients should be reevaluated for response every 2 cycles (6 weeks). Patients who continue on Arm A of treatment for more than 12 months should be reevaluated for response every 3 cycles (9 weeks). In addition to a baseline scan, confirmatory scans should also be obtained 4 weeks following initial documentation of objective response.
Time Frame: after 6 weeks (2 cycles)
Population: Patients that received 2 cycles of treatment. Includes results from patients that crossed over to Arm C.
Measure: Number; unit: participants
Groups:
- Arm A: Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression after 2 cycles of treatment may crossover to arm B.
- Arm C: Crossover From Arm A to B: Cross-over arm: Patients receive oral sorafenib twice daily on days 2-19. Patients also receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A | Arm B | Arm C: Crossover From Arm A to B
Number analyzed (Participants) | 13 | 23 | 5
participants
  Partial Response | 2 | 11 | 1
  Progressive Disease | 8 | 1 | 0
  Stable Disease | 3 | 7 | 4
  Complete Response | 0 | 4 | 0

2. Secondary Outcome: Evaluate the Progression-free Survival Rate
Description: Progression free survival (PFS) was measured by months from the date of treatment to the date of death or the date of progression, and censored at the date of last follow-up for those alive without progression.
Time Frame: up to 85 months of follow-up
Population: Subjects who completed at least 2 cycles of therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Arm C: Crossover From Arm A to B
Number analyzed (Participants) | 13 | 23 | 5
months | 5.6 [3.4 to 17.6] | 16.8 [12.6 to 20.4] | 16.8 [12.6 to 20.4]

3. Secondary Outcome: Overall Survival
Description: Overall survival time, in months, is calculated from the date of treatment to date of death, and to date of last follow-up for those still alive.
Time Frame: up to 85 months of follow-up
Population: Subjects that received at least 2 cycles of treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Arm C: Crossover From Arm A to B
Number analyzed (Participants) | 13 | 23 | 5
months | 25.6 [16.2 to 68.3] | 25.9 [15.4 to 42.1] | 25.9 [15.4 to 42.1]

ADVERSE EVENTS:
Time Frame: Adverse events collected during treatment for all patients over a 7 year period from 2004-2011.
Description: Serious Adverse Event and Adverse Event data reported on Arm A includes events from Arm C patients while on Arm A.
Arm/Group | Arm A | Arm B | Arm C
Serious Adverse Events (participants affected / at risk) | 3/14 | 5/30 | 2/5
Other Adverse Events (participants affected / at risk) | 13/13 | 29/29 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=14) | Arm B (N=30) | Arm C (N=5)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fracture/Right Shoulder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Unrelated to treatment. Patient tripped and fell.
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Keratosis on left lateral forearm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain- Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Secondary Malignancy-Other, excludes metastasis from initial primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased/Neutropenia (Investigations) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=13) | Arm B (N=29) | Arm C (N=5)
Abdominal Bloating (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 7 (9) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 1 (1) | 0 (0)
Alkaline Phosphatase Increase (Investigations) | 2 (2) | 0 (0) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Allergic reaction/hypersensitivity to carboplatin (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (8) | 13 (16) | 2 (2)
Anal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (6) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 5 (13) | 2 (9)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 7 (13) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (7) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (General disorders) | 3 (3) | 4 (4) | 0 (0)
Bleeding gums (Gastrointestinal disorders) | 0 (0) | 1 (6) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (4) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 8 (11) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (16) | 13 (16) | 4 (8)
Dizziness (Nervous system disorders) | 1 (1) | 4 (5) | 0 (0)
Dry Eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 7 (8) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Edema Limbs (General disorders) | 0 (0) | 2 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Fatigue (General disorders) | 8 (20) | 18 (38) | 3 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (2) | 2 (3) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 6 (9) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (8) | 4 (7) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 6 (9) | 12 (19) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (8) | 5 (15) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (10) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 4 (5) | 1 (2)
Infusion Site Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) — Sore throat
Lip Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 0 (0) | 4 (27) | 0 (0)
Mouth Pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Mucosal Infection/Thrush (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 6 (9) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (16) | 0 (0)
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 14 (19) | 2 (4)
Neutrophil count decreased (Investigations) | 2 (7) | 22 (78) | 3 (15)
New right hydroureter (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 0 (0) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (12) | 5 (7) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (14) | 22 (48) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 19 (29) | 3 (8)
Platelet count decreased (Investigations) | 1 (10) | 19 (65) | 3 (13)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (10) | 1 (2)
Rash Pustular (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (22) | 13 (25) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7) | 1 (2)
Scalp Pain (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Karakanthoma on right foot
Stomach Pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 4 (4) | 1 (1)
Vaginal Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge/Yeast Infection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Voice Changes/Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 8 (16) | 0 (0)
Weight Loss (Investigations) | 3 (3) | 2 (3) | 0 (0)
White blood cell decreased (Investigations) | 2 (22) | 15 (71) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less